CLINICAL TRIAL: NCT02876952
Title: Effects of Combined High Intensity Aerobic Interval Training Program and Mediterranean Diet Recommendations in Post-Myocardial Infarct Patients: INTERFARCT Controlled Trial
Brief Title: High Intensity Aerobic Interval Training With Mediterranean Diet Recommendations in Post-Myocardial Infarct Patients
Acronym: INTERFARCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of the Basque Country (UPV/EHU) (Other)
Collaborators: HOSPITAL SANTIAGO APOSTOL. MIRANDA DE EBRO. BURGOS. SPAIN (Unknown)
Responsible Party: Principal Investigator, SARA MALDONADO-MARTIN, PhD Professor, University of the Basque Country (UPV/EHU)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BasqueCU
Record Dates: First submitted 2016-08-07; First posted 2016-08-24 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Myocardial Infarction
Keywords: Cardio-respiratory fitness; high intensity exercise training
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Attention Control Group (AC) (Active Comparator): Moderate to high- intensity physical activity and Mediterranean Diet recommendations
  Interventions: Other: Mediterranean Diet Recommendations; Other: Physical Activity Recommendations
- HV-HIIT (Experimental): Supervised high volume and high intensity interval training exercise group with Mediterranean Diet recommendations.
  High-intensity [heart rate (HR) values up to second ventilatory threshold (VT2) to peak intensity] interval training and high-volume increasing gradually from 20 to 40 min and alternating high and moderate [HR values between first ventilatory threshold (VT1) and VT2] intensities at different protocols.
  Interventions: Other: HIGH VOLUME (HV) Supervised exercise; Other: Mediterranean Diet Recommendations
- LV-HIIT (Experimental): Supervised low volume and high intensity interval training exercise group with Mediterranean Diet recommendations.
  High-intensity (HR values up to VT2 to peak intensity) interval training and low-volume (20 min) alternating high and moderate (HR values between VT1 and VT2) intensities at different protocols.
  Interventions: Other: Mediterranean Diet Recommendations; Other: LOW VOLUME (LW) Supervised exercise

INTERVENTIONS:
Other: HIGH VOLUME (HV) Supervised exercise — Supervised exercise two nonconsecutive days per week (day 1-on the treadmill, day 2-on the bike) for 16 weeks. High-intensity interval training (HIIT) protocol on the treadmill: 5-min warm-up at a moderate-intensity, before walking 2 intervals of 4 min at high-intensity interspersed with intervals of 3 min of walking at moderate-intensity. 1-4 min cool-down at moderate-intensity.
  HIIT protocol on the bike: 5 to 10-min warm-up at moderate intensity. After that, 4 repetitions (1rep = 30 s high-intensity followed by 60 s moderate-intensity) and gradually increased to 16 repetitions in HV-HIIT week by week. 5-10 min cool-down at moderate-intensity
  Arms: HV-HIIT
Other: Mediterranean Diet Recommendations — Participants will be interviewed regarding their usual eating habits. They will receive practical information about which are the Mediterranean Diet (DMed) foods according to the model proposed in the "PREDIMED" trial. Medical doctors or nurses will give this information.
  Before starting the program of intervention, participants will assist to an informative talk in which benefits for the health of the DMed will be exposed and general information about food composition, frequencies of consumption, etc. will be explained.
  Nutritional management: Diet reviews and body mass control will be performed every two weeks to assess the body composition and adherence to treatment. In the event of poor compliance strategies will be addressed for its correction.
Other: Physical Activity Recommendations — Participants will be advised to perform, without supervision, moderate to high-intensity dynamic aerobic exercise (walking, jogging, cycling or swimming) 3-5 days per week, following an adequate warm-up of 5-15 min, at moderate to high intensity (below the ischemic threshold) for a period of 20 to 40 min (not including warm-up and cool-down) followed by a cool-down period of 5-10min. Participants will receive information related to heart rate values regarding moderate and high exercise intensity domains for the self monitoring of exercise intensity.
  Arms: Attention Control Group (AC)
Other: LOW VOLUME (LW) Supervised exercise — Supervised exercise two nonconsecutive days per week (one day on the treadmill, and the second one on the bike) for 16 weeks. HIIT protocol on the treadmill: 5-min warm-up at a moderate-intensity, before walking 2 intervals of 4 min at high-intensity interspersed with intervals of 3 min of walking at moderate-intensity. The training session will end with a 1-4 min cool-down period at moderate-intensity. Total exercise time of 20min HIIT protocol on the bike: 10-min warm-up at moderate intensity. After that, participants will cycle for 4 repetitions (1rep = 30 s high-intensity followed by 60 s moderate-intensity) and gradually increased to 8 repetitions in LV-HIIT week by week. The training session will end with a 5-10 min cool-down period at moderate-intensity.
  Arms: LV-HIIT

SUMMARY:
Acute myocardial infarction (MI) continues remains to be a major cause of death and disability worldwide. Exercise therapy has long been used for rehabilitation purposes and the benefit of regular physical exercise is also well established. The intensity of aerobic exercise training is a key issue in cardiac rehabilitation programmes.Endurance aerobic training is typically performed as continuous training at moderate to-high exercise intensity in steady-state conditions of aerobic energetic yield. However, interval training (i.e., repeated bouts of short-duration, high to severe- or severe to extreme-intensity exercise, separated by brief periods of lower-intensity) has been proposed to be more effective than continuous exercise for improving exercise capacity. Adding to that, health-related adaptations to low-volume and high intensity interval training have been presented.

On the other hand, the Mediterranean Diet has been widely reported to be a model of healthy eating for its contribution to a favourable health status and a better quality of life, reducing in overall mortality from cardiovascular diseases.

Considering all the above mentioned in MI population, the principal objective for the INTERFARCT study will be to assess the effects of different programs of high intensity aerobic interval training and Mediterranean Diet recommendations in the clinical condition, cardio-respiratory fitness, biomarkers, ventricular function and perception of quality of life after myocardial infarction.

Methods/Design: One hundred and fifty people after suffering acute MI will perform different assessments to evaluate clinical history, physical, biochemical and nutritional condition, and quality of life before and after 16-week of follow-up. All participants will receive Mediterranean diet recommendations and will be randomly assigned to attention control group (diet and physical activity recommendations) or exercise groups (diet recommendations plus high-intensity aerobic interval exercise). Participants assigned to an exercise group will train 2 days/week under supervision (day 1-treadmill and day 2-bike protocol). There will be two aerobic exercise groups: 1) high-intensity interval training and high-volume (HV-HIIT) group, and 2) high-intensity interval training and low-volume (LV-HIIT) group.

DETAILED DESCRIPTION:
The management of acute myocardial infarction (MI) continues to undergo major changes, because it remains to be a major cause of death and disability worldwide. Myocardial infarction may be the first manifestation of coronary artery disease or it may occur, repeatedly, in patients with established disease. The term "myocardial infarction" may have major psychological and legal implications for the individual and society. It is an indicator of one of the leading health problems in the world and it is an outcome measure in clinical trials.

Coronary heart disease is a chronic condition and patients are at high risk for new events and premature death. Several evidence-based interventions can improve prognosis. Lifestyle changes should be explained and proposed to the patients before discharge, including cessation of smoking, blood pressure control, and advice regarding diet and weight control, and the encouragement of physical activity. Exercise therapy has long been used for rehabilitation purposes and the benefit of regular physical exercise is also well established. 1 The intensity of aerobic exercise training is a key issue in cardiac rehabilitation programmes. Exercise intensity is directly linked to both the amount of improvement in exercise capacity and the risk of adverse events during exercise, and intensity ranges for aerobic training prescription and design are included in several guidelines and publications regarding secondary prevention and cardiac rehabilitation. Aerobic fitness is recognized as a robust indicator of cardiovascular health and a well-established predictor of total and cardiovascular mortality in subjects with and without coronary heart disease. Direct measurements of peak oxygen uptake (VO2peak) and ventilatory thresholds are considered the gold standard references for the evaluation of aerobic metabolism function and, consequently, for aerobic exercise intensity assessment and design. The increase of VO2peak after a period of exercise training depends of the components of frequency, intensity, time or volume, and type or modality (FITT principle), which constitute the key to achieve a safe exercise training effect. Endurance aerobic training is typically performed as continuous training at moderate to-high exercise intensity in steady-state conditions of aerobic energetic yield. However, interval training (i.e., repeated bouts of short-duration, high to severe- or severe to extreme-intensity exercise, separated by brief periods of lower-intensity) has been proposed to be more effective than continuous exercise for improving exercise capacity. Adding to that, health-related adaptations to low-volume and high intensity interval training have been presented. This type of training is characterized by sessions that involve a relatively small total amount of exercise at high-intensity (i.e., ≤10 min). To our knowledge, there are no studies that compare HIIT with different volume exercise in patients who have suffered MI.

On the other hand, the relevance of overall high-quality food patterns, rather than focus on single nutrients and foods, has emerged as a powerful paradigm to address the diet and to assess their potential cardiovascular disease preventive effects. The Mediterranean Diet, representing the dietary pattern usually consumed among the populations bordering the Mediterranean sea, has been widely reported to be a model of healthy eating for its contribution to a favourable health status and a better quality of life, reducing in overall mortality from cardiovascular diseases.

Considering all the above mentioned in MI population: 1) the combination of the Mediterranean Diet with exercise seems critical in greater reduction of mortality from cardiovascular disease and improved cardiovascular biomarkers, 2) no previous studies have compared the effects of a combined dietary recommendations specific to people after MI with exercise training at high intensity interval training and different volumes (i.e., high- and low-volume).INTERFARCT study is designed to investigate what effect different 16-week aerobic INTERval exercise programs with Mediterranean Diet recommendations will have in people after suffering an acute myocardial inFARCTion.

PRIMARY OBJECTIVE:

To assess the effects of different programs of high intensity aerobic interval training and Mediterranean Diet recommendations in the clinical condition, cardio-respiratory fitness, biomarkers, ventricular function and perception of quality of life after myocardial infarction.

SECONDARY OBJECTIVES

1. To analyze the differences in the studied variables between the two high intensity aerobic interval training programs (high volumen vs low volume) with Mediterranean Diet recommendations to observe the effect of exercise volume.
2. To analyze whether a treatment with only recommendations (exercise and diet) is effective in the secondary prevention of cardiovascular disease comparing to supervised exercise.

ELIGIBILITY:
Inclusion Criteria:

* Two months to 10 years from the cardiovascular event.
* Left ventricular ejection fraction > 30%
* Ability to undertake regular physical activity (walking and biking)

Exclusion Criteria:

* Moderate to severe heart valvular disease.
* Atrial fibrilation.
* Uncontrolled atrial or ventricular arrhythmias.
* Exercise induced myocardial ischaemia.
* Pericardial disease.
* Uncontrolled hypertension.
* Insulin dependent diabetes mellitus.
* Moderate to severe chronic lung disease (Vital capacity and/or forced expiratory volume during the first second <80% to that expected for the age).
* Severe kidney disease (renal creatinine clearance <30 mL/min, calculated by Cockcroft-Gault formula).
* Anaemia (haemoglobin <12 g/dL).
* Life expectancy less than one year.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Direct Cardio-respiratory fitness | 16 weeks
  Direct cardio-respiratory fitness will be evaluated through objectives variables such as peak oxygen uptake and ventilatory thresholds with a cardio pulmonary exercise test.

SECONDARY OUTCOMES:
Left Ventricular Function | 16 weeks
  Left ventricular function will focus on the assessment of cardiovascular hemodynamics by cardiac ultrasound, global cardiac mechanics in systole and diastole, and the relationship between the cardiac structure and regional myocardial function.
Biochemical measures: lipid metabolism | 16 weeks
  Medical doctors will ask for a biochemical analysis including all the below variables to analyze the lipid metabolism of participant:
  Lipid metabolism: total cholesterol (mg/dL), low-density lipoprotein cholesterol (mg/dL), high-density lipoprotein cholesterol (mg/dL), Triglycerides (mg/dL).
Biochemical measures: general metabolism | 16 weeks
  Medical doctors will ask for a general biochemical analysis including all the below variables to analyze a general participant's profile related to:
  General metabolism: urea (mg/dL), creatinine (mg/dL), glomerular filtrate (mL/min), basal glucose (mg/dL), HbA1c (%), insulin, homoeostasis model assessment index (HOMA), uric acid (mg/dL), ionogram, alanine aminotransferase (U/L), aspartate aminotransferase (U/L), blood count.
Biochemical measures: myocardial stress and damage | 16 weeks
  Medical doctors will ask for a general biochemical analysis including all the below variables to analyze a general participant's profile:
  Myocardial damage: troponin T (ng/dL), total and creatine phosphokinase cardiac specific isoenzyme (MB) (U/mL).
  Myocardial stress: brain natriuretic peptide (pg/mL). Neuro-hormonal state: renin, aldosterone (ng/dL). Systemic inflammation: protein C reactive (PCRus) (mg/dL), Interleukin 6 (IL-6) (pg/mL), Tumor necrosis factor-alpha (TNF-alpha) (pg/mL).
  Procoagulant state: D-dimer (ng/mL), fibrinogen (mg/dL). Oxidative stress: ox-LDL (units/mL).
Quality of Life | 16 weeks
  Participants' health-related quality of life will be determined using the 36-item Short Form Medical Outcome Questionnaire (SF-36).
Vascular endothelial function | 16 weeks
  Determination of carotid artery-intima-media thickness through carotid ultrasonography.
Dietary Assessment: dietary recall | 16 weeks
  Dietary intake and habits will be assessed by subjective assessments using open-ended surveys such as dietary recalls or records
Dietary Assessment: food frequency questionnaire | 16 weeks
  Dietary intake and habits will be assessed by subjective assessments using closed-ended surveys including food frequency questionnaires
Dietary Assessment:Mediterranean Diet Adherence Screener questionnaire | 16 weeks
  Dietary intake and habits will be assessed by subjective assessments using Mediterranean Diet Adherence Screener questionnaire.
Height | 16 weeks
  Height (cm)
Body mass | 16 weeks
  body mass (kg)
Waist and hip ratio | 16 weeks
  Measurements:waist and hip perimeters (cm).
Indirect cardiorespiratory fitness | 16-weeks
  Indirect cardiorespiratory fitness will be assessed through a fiel test called Modified Shuttle Walk Test
Assessment of state of depression and anxiety | 16 weeks
  Self-assessment scale instrument for detecting states of depression and anxiety in the setting of an hospital medical outpatient clinic: Hospital Anxiety & Depression Scale
Body composition | 16 weeks
  Bioelectrical impedance analysis (BIA) is a commonly used method for estimating body composition, and in particular body fat, fat free body fat and water. All of them as a percentage of the total body mass

CONTACTS AND LOCATIONS:
Overall Officials: SARA MALDONADO-MARTIN, PhD, Principal Investigator — UNIVERSITY OF THE BASQUE COUNTRY. Department of Physical Education and Sport
Locations (1):
- Department of Physical Education and Sport. Faculty of Education and Sport-Physical Activity and Sport Section. University of the Basque Country, Vitoria-Gasteiz, Araba/álava, Spain

IPD SHARING:
Plan to Share IPD: No
Data won't be shared

REFERENCES:
- [Background] Task Force on the management of ST-segment elevation acute myocardial infarction of the European Society of Cardiology (ESC); Steg PG, James SK, Atar D, Badano LP, Blomstrom-Lundqvist C, Borger MA, Di Mario C, Dickstein K, Ducrocq G, Fernandez-Aviles F, Gershlick AH, Giannuzzi P, Halvorsen S, Huber K, Juni P, Kastrati A, Knuuti J, Lenzen MJ, Mahaffey KW, Valgimigli M, van 't Hof A, Widimsky P, Zahger D. ESC Guidelines for the management of acute myocardial infarction in patients presenting with ST-segment elevation. Eur Heart J. 2012 Oct;33(20):2569-619. doi: 10.1093/eurheartj/ehs215. Epub 2012 Aug 24. No abstract available. PMID 22922416
- [Background] Thygesen K, Alpert JS, Jaffe AS, Simoons ML, Chaitman BR, White HD; Joint ESC/ACCF/AHA/WHF Task Force for the Universal Definition of Myocardial Infarction; Katus HA, Lindahl B, Morrow DA, Clemmensen PM, Johanson P, Hod H, Underwood R, Bax JJ, Bonow RO, Pinto F, Gibbons RJ, Fox KA, Atar D, Newby LK, Galvani M, Hamm CW, Uretsky BF, Steg PG, Wijns W, Bassand JP, Menasche P, Ravkilde J, Ohman EM, Antman EM, Wallentin LC, Armstrong PW, Simoons ML, Januzzi JL, Nieminen MS, Gheorghiade M, Filippatos G, Luepker RV, Fortmann SP, Rosamond WD, Levy D, Wood D, Smith SC, Hu D, Lopez-Sendon JL, Robertson RM, Weaver D, Tendera M, Bove AA, Parkhomenko AN, Vasilieva EJ, Mendis S. Third universal definition of myocardial infarction. Circulation. 2012 Oct 16;126(16):2020-35. doi: 10.1161/CIR.0b013e31826e1058. Epub 2012 Aug 24. No abstract available. PMID 22923432
- [Background] Mezzani A, Hamm LF, Jones AM, McBride PE, Moholdt T, Stone JA, Urhausen A, Williams MA; European Association for Cardiovascular Prevention and Rehabilitation; American Association of Cardiovascular and Pulmonary Rehabilitation; Canadian Association of Cardiac Rehabilitation. Aerobic exercise intensity assessment and prescription in cardiac rehabilitation: a joint position statement of the European Association for Cardiovascular Prevention and Rehabilitation, the American Association of Cardiovascular and Pulmonary Rehabilitation, and the Canadian Association of Cardiac Rehabilitation. J Cardiopulm Rehabil Prev. 2012 Nov-Dec;32(6):327-50. doi: 10.1097/HCR.0b013e3182757050. PMID 23103476
- [Background] Piepoli MF, Corra U, Adamopoulos S, Benzer W, Bjarnason-Wehrens B, Cupples M, Dendale P, Doherty P, Gaita D, Hofer S, McGee H, Mendes M, Niebauer J, Pogosova N, Garcia-Porrero E, Rauch B, Schmid JP, Giannuzzi P. Secondary prevention in the clinical management of patients with cardiovascular diseases. Core components, standards and outcome measures for referral and delivery: a policy statement from the cardiac rehabilitation section of the European Association for Cardiovascular Prevention & Rehabilitation. Endorsed by the Committee for Practice Guidelines of the European Society of Cardiology. Eur J Prev Cardiol. 2014 Jun;21(6):664-81. doi: 10.1177/2047487312449597. Epub 2012 Jun 20. PMID 22718797
- [Background] Piepoli MF, Conraads V, Corra U, Dickstein K, Francis DP, Jaarsma T, McMurray J, Pieske B, Piotrowicz E, Schmid JP, Anker SD, Solal AC, Filippatos GS, Hoes AW, Gielen S, Giannuzzi P, Ponikowski PP. Exercise training in heart failure: from theory to practice. A consensus document of the Heart Failure Association and the European Association for Cardiovascular Prevention and Rehabilitation. Eur J Heart Fail. 2011 Apr;13(4):347-57. doi: 10.1093/eurjhf/hfr017. PMID 21436360
- [Background] Vanhees L, Rauch B, Piepoli M, van Buuren F, Takken T, Borjesson M, Bjarnason-Wehrens B, Doherty P, Dugmore D, Halle M; Writing Group, EACPR. Importance of characteristics and modalities of physical activity and exercise in the management of cardiovascular health in individuals with cardiovascular disease (Part III). Eur J Prev Cardiol. 2012 Dec;19(6):1333-56. doi: 10.1177/2047487312437063. PMID 22637740
- [Background] Guiraud T, Nigam A, Gremeaux V, Meyer P, Juneau M, Bosquet L. High-intensity interval training in cardiac rehabilitation. Sports Med. 2012 Jul 1;42(7):587-605. doi: 10.2165/11631910-000000000-00000. PMID 22694349
- [Background] Gibala MJ, Little JP, Macdonald MJ, Hawley JA. Physiological adaptations to low-volume, high-intensity interval training in health and disease. J Physiol. 2012 Mar 1;590(5):1077-84. doi: 10.1113/jphysiol.2011.224725. Epub 2012 Jan 30. PMID 22289907
- [Background] Martinez-Gonzalez MA, Salas-Salvado J, Estruch R, Corella D, Fito M, Ros E; PREDIMED INVESTIGATORS. Benefits of the Mediterranean Diet: Insights From the PREDIMED Study. Prog Cardiovasc Dis. 2015 Jul-Aug;58(1):50-60. doi: 10.1016/j.pcad.2015.04.003. Epub 2015 May 1. PMID 25940230
- [Background] Sofi F, Cesari F, Abbate R, Gensini GF, Casini A. Adherence to Mediterranean diet and health status: meta-analysis. BMJ. 2008 Sep 11;337:a1344. doi: 10.1136/bmj.a1344. PMID 18786971
- [Derived] Aispuru-Lanche R, Jayo-Montoya JA, Maldonado-Martin S. Vascular-endothelial adaptations following low and high volumes of high-intensity interval training in patients after myocardial infarction. Ther Adv Cardiovasc Dis. 2024 Jan-Dec;18:17539447241286036. doi: 10.1177/17539447241286036. PMID 39380195
- [Derived] Maldonado-Martin S, Jayo-Montoya JA, Matajira-Chia T, Villar-Zabala B, Goiriena JJ, Aispuru GR. Effects of combined high-intensity aerobic interval training program and Mediterranean diet recommendations after myocardial infarction (INTERFARCT Project): study protocol for a randomized controlled trial. Trials. 2018 Mar 2;19(1):156. doi: 10.1186/s13063-018-2529-3. PMID 29499766